CLINICAL TRIAL: NCT02306317
Title: Changing the Paradigm for Improving Neonatal Care: Clinical Study on Optimal Oxygen-saturation Time and the Adding Value of Parents to Nursing Care in the Control of Fi02
Brief Title: The Adding Value of Parents to Nursing Care in the Control of FiO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmen Rosa Pallas (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, Carmen Rosa Pallas, Dra. Carmen Rosa Pallás Alonso, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Neonatología-2014-01
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Premature Birth of Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control by nursing. (Active Comparator): FiO2 adjusted manually by nursing staff. Intervention: Other. Standard procedure
  Interventions: Other: Standard procedure
- Control by parents. (Experimental): FiO2 adjusted manually by parents. Intervention. Other. Experimental procedure
  Interventions: Other: Experimental procedure

INTERVENTIONS:
Other: Standard procedure — FiO2 manually controlled by nursing
  Arms: Control by nursing.
Other: Experimental procedure — FiO2 manually controlled by parents, after training.
  Arms: Control by parents.

SUMMARY:
The purpose of this study is to determine whether saturation control by parents in children younger than 32 weeks or under 1500 g versus conventional care performed by nursing increases the time in which these patients remain at optimal saturation range. If the hypothesis of this study is confirmed premature infants could prevent episodes of hypoxia-hyperoxia and also give more relevance to the role of parents in caring for their children admitted in a neonatal intensive care unit.

DETAILED DESCRIPTION:
Both episodes of hyperoxia and hypoxemia in preterm infants increase morbidity and mortality. Nowadays the adjustment of FiO2 is manually controlled, which means it depends on the staff, needing multiple adjustments throughout the day.

The investigators's hypothesis is that the FiO2 control by parents, improve the percentage of time in range of optimum saturation at least 10% compared to control by nurses.

The aim of this study is to compare the proportion of time with oxygen saturation (SpO2) within the assigned target range, in the preterm infants whose parents modify the fraction of inspired oxygen (FiO2) versus the nursing staff modifying group.

This is a randomized controlled clinical study in the neonatal intensive care unit at Hospital 12 de Octubre. Patients will be randomized in two groups, Experimental Group: parents controlling the saturation ranges, they will manually adjust FiO2 versus the Control Group: controlled by nursing staff (standard procedure). Saturations will be registered and adjustments of FiO2 will be filmed for nonconsecutive 20-hours periods. Twenty-three patients will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Related to child
* Preterm neonates less than 32 weeks or less than 1500 g hospitalized in the Neonatal Intensive Care Unit at Hospital 12 de Octubre.
* Receiving supplemental oxygen ≤0.4 administered by CPAP or conventional nasal cannula or high flow or children with BiPAP (flow generator with double level pressure)
* Minimum age 7 days old.
* Related to the mother:
* Absence of health problems that allows her to perform the task.
* Availability to frequently visit her baby with the father or with a companion, at least for 20 hours, not consecutive.
* Understanding of the study and the Spanish language by the mother and father or companion.
* Signed informed consent.

Exclusion Criteria:

* Evidence of pneumothorax or pneumomediastinum.
* Non-compliance with study protocol.
* Requiring treatment with vasoactive drugs.

Ages: 7 Days to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Children maintained within the saturation ranges in each group | 20-40 hours as maximum
  Percentage of time the child is kept within the ranges of saturation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Carmen R. Pallás Alonso, Dra., Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Pelegrina MD, Lorenzo-Rodriguez A, Lora-Pablos D, Munoz-Amat B, Morales-Betancourt C, Pallas-Alonso CR. FiO2 control by parents of preterm infants admitted to a neonatal intensive care unit: A pilot study. Acta Paediatr. 2018 Aug;107(8):1471-1472. doi: 10.1111/apa.14364. Epub 2018 May 11. No abstract available. PMID 29676033